CLINICAL TRIAL: NCT01973959
Title: Quality of Postoperative Patient Handover in the Post-anaesthesia Care Unit: A Prospective Analysis
Brief Title: Information Transfer During Postoperative Handovers in the Post-anaesthesia Care Unit
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Annika Milby, Postgraduate Student, University of Witten/Herdecke
Other Study IDs: 108/2011; 108/2011 (Other: Ethikkommision der Universität Witten Herdecke)
Record Dates: First submitted 2013-10-21; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Information Transfer During Postoperative Handovers

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anaesthesiology plays a key role in promoting safe perioperative care. This includes the perioperative phase in the post-anaesthesia care unit (PACU) where problems with incomplete information transfer may have a negative impact on patient safety and can lead to patient harm. The objective of this study is to analyse information transfer during postoperative handovers in the PACU.

With a self-developed checklist information transfer during postoperative handovers will be documented and subsequently compared with patient information in anaesthesia records.

ELIGIBILITY:
Inclusion Criteria:

* All patients transferred to the PACU after surgery

Exclusion Criteria:

* Age < 18 years
* patients who have surgery under local anaesthesia or in standby
* patients who are transferred to the surgical intensive care unit (SICU) after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who undergo surgery (general surgery, neurosurgery, ophthalmic surgery, orthopaedics, plastic surgery, trauma surgery, thoracic surgery).
Sampling Method: Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quantity of Information Loss during Postoperative Handovers in the PACU | Two months

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenhaus Köln-Merheim, Departement of Anaesthesiology and Intensive Care Medicine, Cologne, North Rhine-Westphalia, Germany